CLINICAL TRIAL: NCT05603182
Title: A Phase 1, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetics Study of PRA052 in Healthy Volunteers
Brief Title: A Study of PRA052 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prometheus Biosciences, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: PR600-101; MK-8690-001 (Other: Merck)
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAD Cohorts 1-8 Experimental Arm (Experimental): Subjects will receive a single intravenous or subcutaneous dose of PRA052 in a dose escalation format
  Interventions: Drug: PRA052
- SAD Cohorts 1-8 Placebo Arm (Placebo Comparator): Subjects will receive a single intravenous or subcutaneous dose of placebo
  Interventions: Other: Placebo
- MAD Cohorts 1-5 Experimental Arm (Experimental): Subjects will receive three subcutaneous or intravenous doses of PRA052, one dose every 2 weeks, in a dose escalation format
  Interventions: Drug: PRA052
- MAD Cohorts 1-5 Placebo Arm (Placebo Comparator): Subjects will receive three subcutaneous or intravenous doses of placebo, one dose every 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PRA052 — PRA052
  Arms: MAD Cohorts 1-5 Experimental Arm; SAD Cohorts 1-8 Experimental Arm
Other: Placebo — Placebo
  Arms: MAD Cohorts 1-5 Placebo Arm; SAD Cohorts 1-8 Placebo Arm

SUMMARY:
This is randomized, double-blind, placebo-controlled, single and multiple ascending dose study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of PRA052 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (of non-childbearing potential only) between minimum adult legal age (according to local laws for signing the informed consent document) and 60 years of age.
* Male subjects must use reliable forms of contraception during sexual intercourse with female partners from screening to 12 weeks after the end of dosing.
* Good general health as determined by medical history, and by results of physical examination, chest x-ray, vital signs, ECG, and clinical laboratory tests obtained within 28 days (4 weeks) prior to study drug administration

Exclusion Criteria:

* History or presence of any clinically significant organ system disease that could interfere with the objectives of the study or the safety of the subjects.
* Blood pressure and heart rate are outside the ranges 90-140 mmHg systolic, 40-90 mmHg diastolic, heart rate 40-99 beats/min.
* 12-lead ECG with any abnormality judged by the Investigator to be clinically significant, QRS >= 120 milliseconds (msec), or QTcF interval of > 450 msec for men or >470 msec for women.
* Presence or history of any abnormality or illness, which in the opinion of the Investigator may affect absorption, distribution, metabolism or elimination of the study drug.
* Any screening laboratory evaluation outside the laboratory reference range that is judged by the Investigator to be clinically significant.
* History of or current active tuberculosis (TB) infection; history of latent TB that has not been fully treated or current latent TB infection as indicated by a positive QuantiFERON-TB test.
* History of significant allergy to any medication as judged by the Investigator.
* History of alcohol or drug abuse within the past 24 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Up to 20 weeks
  Incidence, severity, and causal relationship of TEAEs

SECONDARY OUTCOMES:
Cmax | Up to 20 weeks
  Maximum concentration after single and multiple ascending doses
Tmax | Up to 20 weeks
  Time to reach maximum concentration after single and multiple ascending doses
t1/2 | Up to 20 weeks
  Half life after single and multiple ascending doses
F% | Up to 20 weeks
  Bioavailability after SC injection
ADA | Up to 20 weeks
  Incidence of anti-drug antibody after single and multiple ascending doses

CONTACTS AND LOCATIONS:
Overall Officials: Prometheus Biosciences, Inc., Study Chair — Prometheus Biosciences, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (1):
- Prometheus Clinical Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/